CLINICAL TRIAL: NCT00867919
Title: Family Therapy for Adolescent Depression: Deployment Focused Development, Phase 1
Brief Title: Designing and Testing a Family Therapy for Adolescent Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH076966 (NIH); R34MH076966 (NIH); DDTR B4-TBI
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive a cognitive behavioral family therapy for adolescent depression to be developed in this study.
  Interventions: Behavioral: Behavioral Family Treatment
- 2 (Active Comparator): Participants will receive treatment as usual 1 year prior to the experimental treatment group.
  Interventions: Other: Community-based treatment as usual

INTERVENTIONS:
Behavioral: Behavioral Family Treatment — 11 to 15 sessions of a cognitive behavioral family therapy that will be developed during the course of this study and will address the following:
  * parent-adolescent conflict
  * adolescent development
  * support and closeness
  * behavioral activation
  * response to adolescent negative affect
  * relapse prevention
  * suicide prevention, if necessary
  Arms: 1
Other: Community-based treatment as usual — Treatment as usual, which will most likely consist of 8 to 10 sessions of community-based depression treatment
  Arms: 2

SUMMARY:
This study will design and test a cognitive behavioral therapy for depressed adolescents that uses family interactions to help with treatment.

DETAILED DESCRIPTION:
Adolescent depression causes persistent feelings of sadness, loss of self-worth, discouragement, and loss of interest in usual activities. Treatments for adolescent depression have mixed success, with 25% to 40% of depressed adolescents still experiencing depressive symptoms at the end of the most effective treatments and gains made in treatment sometimes fading over time. Research suggests that family processes are associated with the effectiveness of treatments for adolescent depression and with reducing symptoms over time. Evidence also shows that treatments developed and tested in a research setting are not easily applied to community settings. This study will first design a cognitive behavioral therapy for adolescent depression that will involve the families of the depressed adolescents and then test the therapy in several settings, including clinics.

Development of this therapy will involve five different groups of participants. Each group will include both depressed adolescents and a parent or guardian. The first group of participants will partake in a focus group, in which they will break into two discussion groups, one of parents and guardians and one of adolescents, that will discuss what kind of help and information would be useful to them and why they would consider seeing a therapist.

The second group will participate in alpha testing, which will involve receiving the first version of the therapy. The therapy is anticipated to include 8 to 12 weekly treatment sessions, with homework assignments to practice their learned skills in everyday life. Participants in alpha testing will also complete interviews and questionnaires at Week 7 and at the end of treatment to assess satisfaction with treatment, treatment clarity, and usefulness of the information and strategies they learned. After alpha testing, the therapy will be revised based on the feedback received. The third group will participate in beta testing, which will involve receiving the second version of the therapy and completing the same assessments as those done by the alpha group.

The fourth group of participants will receive pilot testing of the finalized therapy. This finalized version will involve 11 to 15 weekly sessions. The fifth group will receive treatment as usual from a mental health clinic and serve as a control group to compare to the pilot testing group. Before and after treatment, both of these groups will complete questionnaires and interviews assessing the effectiveness of their treatment and questionnaires and observations of family functioning. All sessions throughout the study involving the newly designed family therapy will be videotaped.

ELIGIBILITY:
Inclusion Criteria:

* Family with an adolescent between 14 and 18 years of age and at least one parent or permanent guardian with whom the adolescent resides
* Family's primary concerns include depressive symptoms
* Adolescent has a score above 24 on the Center for Epidemiological Studies-Depression Scale
* Family will be seeking services at the community mental health center that is associated with the study

Exclusion Criteria:

* Adolescents presenting with evidence of severe difficulties associated with comorbid conditions, such that the focus of treatment would need to shift to nonaffective symptoms
* Adolescents evidencing symptoms of mania or psychoses or with suicidal behaviors requiring inpatient care
* Adolescents with cognitive limitations of severity that will preclude meaningful participation in the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies-Depression (CES-D) Scale | Measured pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa B. Sheeber, PhD, Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - Options Counseling, Eugene, Oregon
  - Oregon Research Institute, Eugene, Oregon